CLINICAL TRIAL: NCT00164710
Title: An Open Randomised Trial of the Efficacy of Sulfadoxine-Pyrimethamine (SP), Amodiaquine + SP (AQ-SP), AQ + Artesunate (AQ-Art), Chlorproguanil-Dapsone + Art (CD-Art), and Lumefantrine-Artemether (LA) for Uncomplicated Malaria in Malawi
Brief Title: Assessing the Efficacy of Four Drug Combinations as the Next First-line Therapy for Uncomplicated Malaria in Malawi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health and Population, Malawi (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-4539; PA# 04018
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Malaria, Falciparum
Keywords: antimalarials
MeSH Terms: conditions — Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; Amodiaquine; Artesunate; chloroguanil, dapsone drug combination; Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine
Drug: amodiaquine plus sulfadoxine-pyrimethamine
Drug: amodiaquine plus artesunate
Drug: chlorproguanil-dapsone plus artesunate
Drug: lumefantrine-artemether

SUMMARY:
Sulfadoxine-pyrimethamine (SP) is the current first-line treatment for uncomplicated malaria in Malawi. The malaria parasite P. falciparum has developed resistance to this drug so that the drug is much less effective than in previous years. This study was developed and conducted in collaboration with the National Malaria Control Programme of Malawi to assess the efficacy of four antimalarial drug combinations to provide evidence to assist the Malawian Ministry of Health in identifying and implementing as policy the next first-line antimalarial for uncomplicated malaria in Malawi. In an open, randomized trial in children under five years of age, four drug combinations, all of which are licensed in Malawi, are being assessed: amodiaquine plus sulfadoxine-pyrimethamine (AQ-SP), amodiaquine plus artesunate (AQ-Art), chlorproguanil-dapsone plus artesunate (CD-Art) and lumefantrine-artemether (LA). SP is also included as a fifth arm of the study for current data on its efficacy. Data on side effects of the drugs will also be collected. The results of this study will provide some of the information necessary to guide the Malawi National Malaria Control Program in selecting its next first antimalarial treatment for uncomplicated malaria. The study adheres to the World Health Organization's 2003 standardized protocol for assessing antimalarial drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 - 59 months
* Axillary temperature ≥ 37.5 °C
* Monoinfection with P. falciparum
* Parasitaemia between 2000 - 200000 parasites/µl
* Haemoglobin concentration (finger-prick blood sample by HemoCue) > 7g/dl
* Consent by the patient's adult guardian
* Residence in the locality and willingness to attend for scheduled visits

Exclusion Criteria:

* altered consciousness
* convulsions
* prostration (inability to sit/stand/suck/drink)
* respiratory distress or breathlessness
* jaundice
* abnormal breathing
* haemoglobinuria
* circulatory collapse
* persistent vomiting (cannot keep down liquids)
* evidence of a diagnosis other than malaria on physical examination
* presence of mixed infection
* presence of severe malnutrition (as evidenced by symmetrical oedema involving at least the feet, light hair color, or cachexia)
* contraindications to the antimalarial drugs used, especially history of allergy
* history of receiving a drug with antimalarial activity in the week prior to enrollment

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 365
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
• Rate of Adequate Clinical and Parasitological Response at 14 days (WHO-defined measure of efficacy)

SECONDARY OUTCOMES:
• Rate of Adequate clinical and parasitological response 28 days
• Mean percent change in blood haemoglobin concentration between day 0 and day 28
• Incidence of adverse events during the period of observation
• Rate of Early Treatment Failure (as defined by the WHO in their 2003 standardized protocol for assessing antimalarial drug efficacy)
• Rate of Late Clinical Failure (as defined by the WHO)
• Rate of Late Parasitologic Failure (as defined by the WHO)
• Percent of patients with a decrease in haemoglobin concentration
• Percent of patients with a decrease in haemoglobin concentration of ≥ 2g/dl
• Prevalence of parasitemia on Day 2
• Prevalence of parasitemia on Day 3
• Gametocyte prevalence on Day 14
• Gametocyte prevalence on Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Bronzan, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- Malawi (3):
  - Kawale Health Center, Lilongwe, Lilongwe District
  - Machinga District Hospital, Liwonde, Machinga District
  - Matiki Health Center, Dwangwa, Nkhotakota District